CLINICAL TRIAL: NCT04880434
Title: A Phase 2 Multicenter Study Evaluating the Efficacy of KTE-X19 in Subjects With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Study of Brexucabtagene Autoleucel (KTE-X19) in Participants With Relapsed/Refractory Mantle Cell Lymphoma (Cohort 3)
Acronym: ZUMA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-102 (Cohort 3); 2015-005008-27 (EudraCT Number)
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — fludarabine; Cyclophosphamide; brexucabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexucabtagene autoleucel (KTE-X19) (Experimental): Participants with relapsed/refractory mantle cell lymphoma will receive conditioning chemotherapy consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day intravenous (IV) infusion for 3 days followed by a single infusion of brexucabtagene autoleucel (KTE-X19) at a targeted dose of 2 x 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg, with a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0 in Cohort 3.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Brexucabtagene autoleucel

INTERVENTIONS:
Drug: Fludarabine — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously
Biological: Brexucabtagene autoleucel — A single infusion of brexucabtagene autoleucel (KTE-X19) anti-CD 19 CAR T cells
  Other Names: KTE-X19; TECARTUS™

SUMMARY:
The goal of this clinical study is to test how well the study drug, brexucabtagene autoleucel (KTE-X19), works in participants with relapsed/refractory (r/r) mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
Study KTE-C19-102 (NCT02601313) enrolled participants with r/r MCL who have been treated with up to 5 prior regimens including a Bruton's tyrosine kinase inhibitor (BTKi) in Cohort 1 and Cohort 2. However, to fulfill FDA Postmarketing Requirement Cohort 3 is added to the study. It will include participants with r/r MCL who have been treated with up to 5 prior regimens but have not received prior therapy with a BTKi.

The primary analysis in Cohort 1 and Cohort 2 is already completed. Data for Cohort 3 will be analyzed separately. Therefore, this separate registration is only for Cohort 3.

After the end of KTE-C19-102, subjects who received an infusion of anti-CD19 CAR T cells will complete the remainder of the 15-year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Key Inclusion Criteria:

* Up to 5 prior regimens for MCL. Prior therapy must have included anthracycline- or bendamustine-containing chemotherapy and anti-CD20 monoclonal antibody therapy. Individuals must not have received prior therapy with a BTKi.
* At least 1 measurable lesion
* Platelet count ≥ 75,000/uL
* Creatinine clearance (as estimated by Cockcroft Gault) ≥ to 60 cc/min
* Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA), and no clinically significant electrocardiogram (ECG) findings
* Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria:

* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive). Individuals with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing
* History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with central nervous system (CNS) involvement
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per Lugano Classification as Determined by the Independent Radiology Review Committee (IRRC) | Up to 4 years
  ORR is defined as the incidence of either a complete response (CR) or partial response (PR) per the Lugano Classification as determined by IRRC.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 4 years
  DOR is defined as the time from their first objective response to disease progression or death.
Percentage of Participants With Best Objective Response (BOR) | Up to 4 years
  Best objective response is defined as the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable as best response to treatment.
Objective Response Rate (ORR) per Lugano Classification as Determined by Investigators | Up to 4 years
  ORR, as determined by investigators, is defined as the incidence of either a complete response (CR) or partial response (PR) per the Lugano Classification.
Progression Free Survival (PFS) | Up to 4 years
Overall Survival | Up to 4 years
Percentage of Participants Experiencing Treatment-Emergent Adverse Events | Up to 4 years
Percentage of Participants With Clinically Significant Changes in Laboratory Values | Up to 4 years
Percentage of Participants Who Develop Anti-CD19 CAR Antibodies | Up to 4 years
Levels of Anti-CD19 CAR T Cells in Blood | Up to 4 years
Levels of Cytokines in Serum | Up to 4 years
Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Scale Score | Baseline and up to 24 months
  The European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each dimension the participant is asked for a three-level assessment of their health on the current day: "no problems" (1), "some problems" (2), "extreme problems" (3). EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 (worst health state) to 1.00 (perfect health state). Positive numbers indicate improvement from baseline.
Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Visual Analogue Scale (VAS) Score | Baseline and up to 24 months
  EQ-5D is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-consists of two components: a health state profile and an optional visual analogue scale (VAS). The EQ5D-VAS records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. EQ-5D-VAS: range 0 to 100. A higher score indicates better self-reported health status.
Changes in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) Score from Baseline Over Time | Baseline and up to 6 months
  EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions use 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores are averaged, transformed to 0-100 scale; higher score indicate high QoL. A positive change from baseline indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (40):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Stanford University, Palo Alto, California
  - University California Los Angeles (UCLA), Santa Monica, California
  - Sarah Cannon- Denver, Denver, Colorado
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Aurora Health - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon - Tenessee, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Cancer Hospital, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- France (5):
  - CHU de Montpellier, Montpellier
  - Hospital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes, Rennes
- Germany (3):
  - Johannes Gutenberg University Hospital-University Mainz, Mainz
  - Munich University of Technology-Medical Faculty- Ethics Committee, München
  - Universitaetsklinikum Wuerzburg, Würzburg
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam
- Spain (3):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - Queen Elizabeth University Hospital, Glasgow
  - Kings College Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Meerten T, Kersten MJ, Iacoboni G, Hess GR, Mutsaers PGNJ, Martin Garcia-Sancho AM, Goy A, Gine E, Hill BT, Weng WK, Reagan PM, Patel K, Galal A, Herbaux C, Sanderson R, Forcade E, Topp MS, Houot R, Zheng D, Zhang W, Kanska J, Shen RR, Damico Khalid R, Kloos I, Dreyling M, Wang ML. Brexucabtagene autoleucel for BTKi-naive relapsed/refractory mantle cell lymphoma: primary analysis of ZUMA-2 Cohort 3. Blood. 2025 Oct 29:blood.2025029734. doi: 10.1182/blood.2025029734. Online ahead of print. PMID 41160777
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-102%20(Cohort%203)